CLINICAL TRIAL: NCT02846597
Title: Sustained Lung Inflation at Birth for Preterm Infants at Risk of Respiratory Distress Syndrome: the Proper Pressure and Duration: Prospective Randomized Study
Brief Title: Proper Pressure and Duration of Sustained Lung Inflation in Preterm Infants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mansoura University Children Hospital (Other)
Responsible Party: Principal Investigator, Nehad Nasef, Associate Professor, Mansoura University Children Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NICU MUCH 2016
Record Dates: First submitted 2016-07-22; First posted 2016-07-27 (Estimated); Last update posted 2018-04-03 (Actual); Status verified 2018-04

CONDITIONS: Respiratory Distress Syndrome
Keywords: Respiratory distress syndrome; Sustained lung inflation; Delivery room
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Control (No Intervention): Infants in this group will not receive sustained lung inflation in the delivery room and will be put immediately on CPAP at a pressure of 5 cm H2O.
- High pressure for long duration (Active Comparator): Infants in this group will receive sustained lung inflation in the delivery room at a pressure of 20 cm H2O for a duration of 20 second for a single intervention followed by CPAP at a pressure of 5 cm H2O.
  Interventions: Procedure: Sustained lung inflation in preterms (SLI).
- High pressure for short duration (Active Comparator): Infants in this group will receive sustained lung inflation in the delivery room at a pressure of 20 cm H2O for a duration of 10 second for a single intervention followed by CPAP at a pressure of 5 cm H2O.
  Interventions: Procedure: Sustained lung inflation in preterms (SLI).
- Low pressure for long duration (Active Comparator): Infants in this group will receive sustained lung inflation in the delivery room at a pressure of 15 cm H2O for a duration of 20 second for a single intervention followed by CPAP at a pressure of 5 cm H2O.
  Interventions: Procedure: Sustained lung inflation in preterms (SLI).
- Low pressure for short duration (Active Comparator): Infants in this group will receive sustained lung inflation in the delivery room at a pressure of 15 cm H2O for a duration of 10 second for a single intervention followed by CPAP at a pressure of 5 cm H2O.
  Interventions: Procedure: Sustained lung inflation in preterms (SLI).

INTERVENTIONS:
Procedure: Sustained lung inflation in preterms (SLI). — Providing a positive pulmonary ventilation with an opening lung pressure for the first breath of preterm infant for a sustained period of time
  Arms: High pressure for long duration; High pressure for short duration; Low pressure for long duration; Low pressure for short duration

SUMMARY:
The appropriate pressure and duration needed for sustained lung inflation in preterm infants at risk of respiratory distress syndrome have not been well evaluated. We aim for evaluating two different pressures, 20 and 15 cm H2O, for two different duration, 10 and 20 seconds, during the application of sustained lung inflation in the resuscitation of preterm infants with respiratory distress in the delivery room.

DETAILED DESCRIPTION:
This study will be a randomized prospective pilot study in Mansoura University Hospital then the cases were followed at Neonatal Intensive Care Unit in Mansoura University Children Hospital, Mansoura, Egypt.

Preterm infants born equal to or less than 32 weeks gestation with respiratory distress syndrome will be included in the study.

We aim to study the proper pressure and duration of sustained lung inflation in the delivery room.

Preterm infants will be divided into 5 groups:

1. Group 1 (Control group). In this group preterm infants will not be treated with sustained lung inflation and in stead will receive regular respiratory care
2. Group 2 (High pressure for long duration group). Preterm infants in this group will be treated with sustained lung inflation at pressure of 20 cm H2O for 20 seconds
3. Group 3 (High pressure for short duration group). Preterm infants in this group will be treated with sustained lung inflation at pressure of 20 cm H2O for 10 seconds.
4. Group 4 (Low pressure for long duration group). Preterm infants in this group will be treated with sustained lung inflation at pressure of 15 cm H2O for 20 seconds.
5. Group 5 (Low pressure for short duration group). Preterm infants in this group will be treated with sustained lung inflation at pressure of 15 cm H2O for 10 seconds

Sustained lung inflation will be delivered using the T - piece ventilator (Neopuff infant resuscitator; Fisher & Paykel, Auckland, New Zealand ).

All preterm infants with respiratory distress will follow the following steps for neonatal resuscitation

1. All infants will receive initial care including providing warmth, clearing the airway, and drying and stimulating the infant.
2. After the initial steps, pulse oximetry will be initiated to determine oxygen saturation and to guide the required FIO2.
3. Infants in the intervention groups will receive a single single maneuver of sustained lung inflation with the first breath according to the study group.
4. Continuous positive airway pressure at a pressure of 5 cm H2O and FIO2 of 30% will be delivered to infants in the control group immediately after initial steps of resuscitation and to all infants in the intervention groups after the single maneuver of sustained lung inflation.
5. Positive pressure ventilation will be provided uring the T-piece resuscitator if the infant has an inadequate respiratory effort or a heart rate <100 beats per minute at a rate of 40 to 60 times per minute for 30 seconds, after which the heart rate is measured.
6. Oxygen therapy will be titrated to keep a pre-ductal saturation between 90-95%.
7. Endotracheal intubation will be provided if positive pressure ventilation is ineffective, prolonged apnea, or chest compression is required.
8. Chest compression will be required if the infant's heart rate remains <60 bpm despite adequate ventilation for 30 seconds.
9. Surfactant will be administered to preterm infants requiring a fraction of inspired oxygen of 40 percent or higher to maintain oxygen saturation above 90 percent or remain apneic.
10. Mechanical ventilation will be initiated for preterm infants with respiratory acidosis documented by an arterial pH <7.2 and PaCO2 >60 to 65 mmHg, hypoxia documented by an arterial PaO2 <50 mmHg despite FiO2 exceeds 40 percent on nasal continuous positive airway pressure, or severe apnea.

The primary outcome of the study will be the need for endotracheal intubation in the delivery room.

Secondary outcomes include the need for surfactant therapy, the need for endotracheal intubation and mechanical ventilation within 72 hours of birth, the duration of mechanical ventilation and oxygen support, development of air leak syndromes, length of hospital stay, bronchopulmonary dysplasia, necrotising enterocolitis, intraventricular haemorrhage, retinopathy of prematurity, and neonatal mortality before hospital discharge,.

Broncho alveolar lavage will be performed to endotracheally intubated infants enrolled in this study to measure the level of IL-10 as a lung inflammatory marker immediately after birth (basal) then 12 hours after birth (follow up).

ELIGIBILITY:
Inclusion Criteria:

Preterm infants with gestational age ≤ 32 weeks' gestation, presented with respiratory distress syndrome at birth

Exclusion Criteria:

1. - Preterm infants with no manifestations of respiratory distress syndrome at birth.
2. - Presence of major congenital malformation (dysmorphic features or anomalies incompatible with life) .

Ages: 1 Day to 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2013-03; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
The need for endotracheal intubation in the delivery room | One hour

SECONDARY OUTCOMES:
The need for mechanical ventilation | 72 hours
Need of surfactant | 72 hours
Neonatal mortality | 90 days
  Death before hospital discharge
Broncho Pulmonary Dysplasia ( BPD ) | 90 days
  Requirement for oxygen therapy more than 30% by 36 weeks corrected gestational age
Intra-Ventricular Hemorrhage ( IVH ) | 14 days
Retinopathy of Prematurity ( ROP ) | 50 days
Necrotizing Entero Colitis ( NEC ) | 40 days
Length of neonatal intensive care ( NICU ) and hospital stay | 90 days
Air-leak syndrome | 14 days
  Development of pneumothorax or pneumomediastinum

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University Children Hospital, Al Mansurah, El Dakahlya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided